CLINICAL TRIAL: NCT06359262
Title: Feasibility, Effectiveness and Overall Impact of the Hope@School Universal Prevention Program Promoting Child and Adolescent Mental Health in Schools: A Two-arm Randomized Controlled Trial Across Seven European Countries
Brief Title: Evaluating the Hope@School Prevention Program
Acronym: Hope@School
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jens Högström, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KI-HAS-001
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Wellness 1
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hope@School (Experimental): The universal prevention program Hope@School. A digital platform with a number of tools that target mental health and wellbeing in children and adolescents.
  Interventions: Other: Hope@School
- Treatment as usual (Active Comparator): Regular student health care in the schools
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Hope@School — A digital platform aimed at promoting student mental health in schools
  Arms: Hope@School
Other: Treatment as usual — Regular student health care in schools
  Arms: Treatment as usual

SUMMARY:
This multi-center cluster-randomized controlled trial aims to evaluate the feasibility, effectiveness and overall impact of the Hope@School (H@S) program by comparing mental health outcomes in students participating in the H@S program with students having only access to regular student health care (treatment as usual - TAU).

The primary objectives of the study are:

To determine if the H@S program is feasible, acceptable, usable and safe for students, families, teachers and school leaders To establish if the H@S program is associated with improvements in quality of life, everyday functioning, peer relations and general mental health.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 18 years
* Attends school included in the study
* Consents to participate

Exclusion Criteria:

- Younger than 8 and older than 18 years

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3220 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
KIDSCREEN-27 Child version | Baseline, 3 month and 6 month (the 6 month assessment is the primary endpoint)
  Level of child-rated quality of life as measured by a questionnaire

SECONDARY OUTCOMES:
KIDSCREEN-27 Parent version | Baseline, 3 month and 6 month (the 6 month assessment is the primary endpoint)
  Level of parent-rated quality of life (the child's quality of life) as measured by a questionnaire
Mental Health-Promoting Knowledge (MHPK-10) | Baseline, 3 month and 6 month (the 6 month assessment is the primary endpoint)
  Level of child-rated mental health literacy as measured by a questionnaire
Healthy Behaviours in School-aged Children survey protocol (HBSC) part 1 | Baseline, 3 month and 6 month (the 6 month assessment is the primary endpoint)
  Level of child-rated healthy behaviours as measured by a questionnaire
Digital Addiction Scale for Children (DASC) | Baseline, 3 month and 6 month (the 6 month assessment is the primary endpoint)
  Level of child-rated addictive digital behaviours as measured by a questionnaire
Healthy Behaviours in School-aged Children survey protocol (HBSC) part 2 | Baseline, 3 month and 6 month (the 6 month assessment is the primary endpoint)
  Level of child-rated harmful digital practices as measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jens Högström, Ass prof, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided